CLINICAL TRIAL: NCT00892086
Title: Prevalence and Recognition of Geriatric Syndrome in Outpatient Clinic at Srinagarind Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Dr Watchara Boonsawat, Faculty of medicine, Khon Kaen University, Khon Kaen , Thailand
Other Study IDs: I52109
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Dementia; Cognitive Impairment; Depression; Urinary Incontinence; Constipation; Falls
Keywords: geriatric syndrome; immobility
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Depression; Urinary Incontinence; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect the prevalence of geriatric syndrome, which is recognized by an internist, and to compare the data based on the comprehensive geriatric assessment by a geriatrician. The secondary outcome is to develop a practical collected form for the internist.

ELIGIBILITY:
Inclusion Criteria:

* all patients who are over than 60 years old who visit internal medicine outpatient clinic

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: internal medicine outpatient clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-01 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Comparing the prevalence of geriatric syndrome between internist and geriatrician | 1 year

SECONDARY OUTCOMES:
Development of a practical form to collect patient's data | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Srinagarind hospital, Khon Kaen university, Muang District, Changwat Khon Kaen, Thailand